CLINICAL TRIAL: NCT06650917
Title: Explore the Application Effect of Acupoint Massage Combined With Ear Point Pressing Beans in the Remission Stage of Asthma
Brief Title: Acupoint Massage Combined With Ear Point Pressing Beans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hai'an Hospital of TCM001 (Other)
Responsible Party: Principal Investigator, Xiaohong Chu, Deputy Chief Chinese Medicine Practitioner, Hai'an Hospital of TCM001
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hai'an Hospital of TCM001
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental)
  Interventions: Behavioral: the experiment group were treated acupoint massage combined with ear point pressing beans
- control group (Active Comparator)
  Interventions: Behavioral: the control group were treated with acupoint massage

INTERVENTIONS:
Behavioral: the experiment group were treated acupoint massage combined with ear point pressing beans — Salmeterol Xinafoate and Fluticasone Propionate Powder for Inhalation was used 1 puff each time, 2 times/d.
  Patients in the experiment group were treated with auricular point pressing on basis if the treatment of the control group. Selecting 10 acupoints including Tanzhong, Tiantu, Dingchuan(both sides), Feishu(both sides), Yuji(both sides), and Lieque(both sides), and massage each acupoint for about 3 minutes. Acupoint massage once a day from Monday to Friday, lasting for 30 minutes each time. Selecting the Fengxi(both sides), Lung(both sides), Bronchial(both sides), and Shenmen(both sides) acupoints on the ear for ear point pressing beans. The operator rubs the above acupoints with their hands for about 5 minutes, and then performs ear point pressing beans on these 4 acupoints. The ear point pressing beans is performed once a day from Monday to Friday.
  Arms: experiment group
Behavioral: the control group were treated with acupoint massage — Salmeterol Xinafoate and Fluticasone Propionate Powder for Inhalation was used 1 puff each time, 2 times/d.
  On this basis, patients in the control group were treated with acupoint massage.
  Arms: control group

SUMMARY:
Objective: To explore the application effect of acupoint massage combined with ear point pressing beans in the remission stage of asthma. Methods: 120 children with asthma in remission who were treated in pediatric outpatient department from January 2016 to October 2022 were randomly divided into experimental group and control group, with 60 cases in each group.The patients in both groups were treated with salmeterol and fluticasone inhalation powder once a day, twice a day. The patients in the control group were treated with acupoint massage on this basis. Acupoint massage once a day from Monday to Friday, lasting for 30 minutes each time.The patients in the experimental group were treated with ear point pressing beans on the basis of the control group. The ear point pressing beans is performed once a day from Monday to Friday. Changes in pulmonary function and asthma control were observed before and after treatment in the two groups were observed, and forced expiratory volume 1 second (FEV1),forced expiratory vital capacity (FVC), FEV1/FVC, asthma control test scale (ACT) score were compared.

ELIGIBILITY:
Inclusion Criteria:

* The patient met the diagnostic criteria of asthma remission in the Guidelines for prevention and treatment of bronchial asthma；
* 1~18 years old, course of disease > 1 year;
* Patients with complete clinical data and able to cooperate with treatment.

Exclusion Criteria:

* Patients with other cardiopulmonary system diseases or myasthenia gravis;
* Eczema, ulcer or other symptoms in the auricle or skin;
* Illiteracy, cognitive, language or communication disorders;
* The patient has taken medication for asthma treatment within 3 months.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 1 minutes
  Forced expiratory vital capacity (FVC), FEV 1 and FEV1/FVC ratio were measured with Jaeger pulmonary function testing instrument
Asthma control | 1 hour
  The Asthma Control test Scale (ACT) was used for assessment, including daily life status, dyspnea times, asthma symptoms, emergency medication use, and asthma control. Each item was 1 to 5 points, and the total score was 5 to 25 points.
Efficacy assessment | 1 hour
  Complete control: no symptoms occurred throughout the day after treatment, no significant limitation of activity, no acute attack, PEF or FEV1 normal value or ≥ normal expected value; Partial control: after treatment, symptoms> 2 times/week during the day, wake up at night, mild limitation of activity. Drug relief is required for over 2 times/week; Uncontrolled: frequent symptoms during the day and at night, limited activity, acute attacks. Drugs should be used frequently for relief. Total control rate = complete control rate + partial control rate.

IPD SHARING:
Plan to Share IPD: No